CLINICAL TRIAL: NCT03611777
Title: Non-interventional, Cross-sectional, Multicenter Study to Describe the Exacerbations Profile of COPD Patients Treated With ICS in a Real-life Primary Care Population in Spain. OPTI Study.
Brief Title: The OPTI Study in Spain Looks at the History Flare-ups in Patients With Chronic Obstructive Pulmonary Disease (COPD) Treated With Inhaled Steroids.
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237-0070
Record Dates: First submitted 2018-07-02; First posted 2018-08-02 (Actual); Results first posted 2021-02-17 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- subjects with Pulmonary Disease, Chronic Obstructive
  Interventions: Drug: Inhaled corticosteroid

INTERVENTIONS:
Drug: Inhaled corticosteroid — Drug

SUMMARY:
This non-Interventional, descriptive, cross-sectional cohort and multicentre study will be conducted with COPD patients attended at Spanish Primary Care offices.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to participation
2. Female and male patient ≥ 40 years of age
3. Chronic Obstructive Pulmonary Disease (COPD) diagnosis more than 2 years before the study visit
4. Previously confirmed Chronic Obstructive Pulmonary Disease (COPD) diagnosis (post-bronchodilator FEV1/FVC ratio <70%)
5. Clinical data available 2 years before the study visit
6. Ability to complete CAT - COPD Assessment Test

Exclusion Criteria:

1. Current participation in any clinical trial involving a drug or device
2. A moderate or severe exacerbation (requiring oral corticosteroid, antibiotics or hospitalisation) during the study visit or within 4 weeks before the study visit

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: study will be conducted with COPD patients attended at Spanish Primary Care offices.
Sampling Method: Non-Probability Sample
Enrollment: 901 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mireia Canals, (+34) 93 404 58 77, Study Chair — mireia.canals@boehringer-ingelheim.com
Locations (169):
- Spain (169):
  - CS A Pontenova, A Pontenova, Lugo
  - CAP Abrera, Abrera, Barcelona
  - CS Zona VI, Albacete
  - CS Zona IV, Albacete
  - CS Nuestra Señora de la Oliva, Alcalá de Guadaira, Sevilla
  - EAP Carmen Calzado, Alcalá de Henares, Madrid
  - CS Alcasser, Alcasser, Valencia
  - CS La Chopera, Alcobendas, Madrid
  - CS Algeciras Norte, Algeciras, Cádiz
  - CS Algemesi, Algemesi, Valencia
  - CS Almonte, Almonte, Huelva
  - Consultorio Alpuente, Alpuente, Valencia
  - CS Argamasilla de Calatrava, Argamasilla de Calatrava, Ciudad Real
  - CS Baltar Sanxenxo, Baltar, Pontevedra
  - Consultorio Bañaderos, Bañaderos, Las Palmas
  - CAP Sant Marti (EAP Verneda Nord), Barcelona
  - CAP Sants, Barcelona
  - EAP Vía Roma, Barcelona
  - CAP Casernes, Barcelona
  - CAP Chafarinas, Barcelona
  - CAP Trinitat Vella, Barcelona
  - Cap Sant Rafael, Barcelona
  - CAP Casanova, Barcelona
  - CAP Dr. Carles Ribas, Barcelona
  - EAP Guinardo, Barcelona
  - CS Bedman, Bedman, Jaén
  - Consultorio Médico Begíjar, Begíjar, Jaén
  - CS Benigánim, Benigánim, Valencia
  - C. S. Benimamet, Benimamet, Valencia
  - CS Santutxu, Bilbao
  - CS Comuneros, Burgos
  - CS Gamonal Antigua, Burgos
  - CS Matrona Antonia Mesa Fernández, Cabra, Córdoba
  - CS Olivillo, Cadiz
  - C.S. Callosa del Segura, Callosa de Segura, Alicante
  - C.S. Carballo, Carballo, A Coruña
  - CS Nuestra señora de Gracia, Carmona, Sevilla
  - CS Cartaya, Cartaya, Huelva
  - C.S. San Agustín, Castellon
  - CS Catarroja, Catarroja, Valencia
  - CAP Canaletas, Cerdanyola, Barcelona
  - CS Chapela, Chapela, Pontevedra
  - CS Ciudad Rodrigo, Ciudad Rodrigo Salamanca
  - CS Collado Villalba Estación, Collado Villalba, Madrid
  - CS Virgen de la Estrella 2, Coria Del Río, Sevilla
  - CS Jaime Vera, Coslada, Madrid
  - CS Cuenca IV, Cuenca
  - C.S. Cuntis, Cuntis, Pontevedra
  - Consultorio Guargacho, El Monte, Tenerife
  - CS Puerto de Santa María Sur, El Puerto de Santa María, Cádiz
  - CS San Miguel Basauri, Elexalde, Bizcaia
  - CAP Pubilla Casas, Esplugues de Llobregat, Barcelona
  - CS Lobillas, Estepona, Málaga
  - CS Favara, Favara, Valencia
  - CAP Figueres Ernest Lluch, Figueres, Girona
  - CAP Josep Masdevall, Figueres, Girona
  - CS Panaderas, Fuenlabrada, Madrid
  - CS Cuzco, Fuenlabrada, Madrid
  - CS Natahoyo, Gijón
  - CAP Montilivi, Girona
  - Consultorio Gorraiz, Gorráiz
  - CAP Hostalric, Hostalric, Girona
  - CS Huelva Centro, Huelva
  - CS Bulevar, Jaén
  - C.S. Jávea, Jávea, Alicante
  - EAP - Centre - L´Hospitalet de Llobregat, L'Hospitalet de Llobregat, Barcelona
  - CAP Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - CS La Almunia de Doña Godina, La Almunia de Doña Godina, Zaragoza
  - CS La Bañeza II, La Bañeza, León
  - CS La Cañada, La Cañada, Almería
  - CS La Carlota, La Carlota, Córdoba
  - CS La Línea Poniente, La Línea de La Concepción, Cádiz
  - CS La Roda, La Roda, Albacete
  - CS Zubia, La Zubia, Granada
  - CS Laredo, Laredo, Cantabria
  - CS Las Cabezas de San Juan, Las Cabezas, Sevilla
  - CS San José, Las Palmas
  - CS Maspalomas, Las Palmas
  - CS Eras de Renueva, León
  - CS Loeches, Loeches, Madrid
  - CS Lora del Río Virgen de Setefilla, Lora Del Río, Sevilla
  - CS Los Barrios, Los Barrios, Cádiz
  - CS Lucena, Lucena, Córdoba
  - CS San Roque, Lugo
  - CS Montesa, Madrid
  - CS Goya, Madrid
  - CS Potosí, Madrid
  - CS Alcalá de Guadaira, Madrid
  - CS Abrantes, Madrid
  - CS Canal de Panamá, Madrid
  - CS Estrecho de Corea, Madrid
  - CS Arroyo Media Legua, Madrid
  - CS Villa de Vallecas, Madrid
  - CS Aquitania, Madrid
  - CS Villaamil, Madrid
  - CS General Fanjul, Madrid
  - CS Las Aguilas, Madrid
  - CS Entrevias, Madrid
  - CS Malagon, Malagon, Ciudad Real
  - CS Son Rullan, Mallorca
  - CS Mansilla de las Mulas, Mansilla de Las Mulas, León
  - C.M. Mataró, Mataró
  - CS Huelin, Málaga
  - CS Victoria, Málaga
  - CS Meliana, Meliana, Valencia
  - CS Mengibar, Mengibar, Jaén
  - CS Moguer, Moguer Huelva
  - CS Montoro, Montoro, Córdoba
  - CS dos de Mayo, Móstoles, Madrid
  - CS Dr. Luengo Rodríguez, Móstoles, Madrid
  - CS Neda, Neda, Coruña
  - CS Novelda, Novelda, Alicante
  - CS Orgiva, Orgiva, Granada
  - C.S. Osuna, Osuna, Sevilla
  - CS Jardinillos, Palencia
  - CS La Puebla, Palencia
  - CS Pintor Oliva, Palencia
  - CS Palos de la Frontera, Palos de La Frontera, Huelva
  - C.S. Parador, Parador de Las Hortichuelas, Almería
  - C. S. Paterna, Paterna, Valencia
  - CS Pedralba, Pedralba, Valencia
  - Consultorio Peñíscola, Peñíscola, Castellón
  - CS Pilas, Pilas, Sevilla
  - CS Polinya de Xuquer, Polinya de Xuquer, Valencia
  - CS Port de Pollença, Pollença, Baleares
  - CS Lérez, Pontevedra
  - CS Repelega, Portugalete, Bizkaia
  - CS Castaños, Portugalete, Vizcaya
  - CS Puebla de Cazalla, Puebla de Cazalla, Sevilla
  - CS Puerto Lumbreras, Puerto Lumbreras, Murcia
  - CS Puertollano I, Puertollano, Ciudad Real
  - CS Rute, Rute, Córdoba
  - CS Periurbana Sur, Salamanca
  - CS La Cuesta, San Cristóbal La Laguna, Tenerife
  - CS San Fernando Dr. Cayetano Roldán, San Fernando, Cádiz
  - C. S. San Juan, San Juán de Alicante
  - CS Sancti Spiritus, Sancti Spiritus, Salamanca
  - CS Sangüesa, Sangüesa, Navarra
  - CAP Montclar, Sant Boi de Llobregat, Barcelona
  - CAP Dr. Vilaseca, Santa Coloma Gramanet, Barcelona
  - CS San Miguel de Abona, Santa Cruz de Tenerife
  - CS El Doctoral, Santa Lucía de Tirajana, Las Palmas
  - CS Santa María del Camí, Santa Mª Del Camí, Baleares
  - CS Perello, Sueca, Valencia
  - CS Sueca, Sueca, Valencia
  - CS Tacoronte, Tacoronte, Tenerife
  - CS Titaguas, Titaguas, Valencia
  - CS Torredelcampo, Torre Del Campo, Jaén
  - CS Brújula, Torrejón de Ardoz Madrid
  - CS Covadonga, Torrelavega, Cantabria
  - CS Carihuela, Torremolinos
  - CS Tudela Este, Tudela, Navarra
  - CS Valdefuentes, Valdefuentes, Cáceres
  - CS Ingeniero Joaquim Benlloch, Valencia
  - C.S. Malvarrosa, Valencia
  - CS Barrio de la Luz, Valencia
  - CS Campanar, Valencia
  - CS Vélez Norte, Vélez-Málaga
  - CS La Doblada, Vigo
  - C.S. Coia Vigo, Vigo
  - C. S. Almassera de Tonda, Vila Joiosa, Vila Joiosa, Alicante
  - CAP María Bernades, Viladecans, Barcelona
  - C. S. Xunqueira de Ambia, Xunqueira de Ambia, Ourense
  - CS Seminario, Zagaroza
  - CS Virgen de la Concha, Zamora
  - CS Fuentes Norte, Zaragoza
  - CS Canal Imperial Venecia, Zaragoza
  - CS Casablanca, Zaragoza
  - CS Seminario, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions: 1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).Requestors can use the following link http://trials.boehringer-ingelheim.com/ to:
  1. find information in order to request access to clinical study data, for listed studies.
  2. request access to clinical study documents that meet criteria, and upon a signed 'Document Sharing Agreement'

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Non-interventional, cross-sectional, multicenter study to describe the chronic obstructive pulmonary disease (COPD) patient profile of patients treated with or without Inhaled CorticoSteroids (ICS) in primary care, in Spain.
Pre-assignment Details: Only subjects that met all the study inclusion and none of the exclusion criteria were to be entered in the study.
Groups:
- COPD Patients Treated With ICS at Study Visit: Patients with chronic obstructive pulmonary disease (COPD) currently (at study visit) treated with Inhaled CorticoSteroids (ICS).
- COPD Patients Not Treated With ICS at Study Visit: Patients with chronic obstructive pulmonary disease (COPD) currently (at study visit) not treated with Inhaled CorticoSteroids (ICS).
Period: Overall Study
Arm/Group | COPD Patients Treated With ICS at Study Visit | COPD Patients Not Treated With ICS at Study Visit
Started | 432 | 469
Completed | 432 | 469
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): Patients who provided informed consent and fulfilled all selection criteria, totalled 901 patients. Of those, 545 patients received at least one dose of ICS during 2 years prior to the study period. Further, a total of 441 patients were considered for the safety analysis related to a BI product, including those patients receiving Spiolto®, Striverdi®, Spiriva®, Atrovent® during the study period.
Groups:
- Total: Total of all reporting groups
Arm/Group | COPD Patients Treated With ICS at Study Visit | COPD Patients Not Treated With ICS at Study Visit | Total
Number analyzed (Participants) | 432 | 469 | 901
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.44 (10.27) | 70.55 (9.37) | 70.97 (9.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 88 | 177
  Male | 343 | 381 | 724
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 427 | 467 | 894
  African | 3 | 1 | 4
  Argentinian | 0 | 1 | 1
  Gypsy | 1 | 0 | 1
  Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Currently on Inhaled CorticoSteroids (ICS) Who Did Not Have Moderate or Severe Exacerbation in the Year Prior to the Study Visit
Description: Percentage of patients currently on ICS who did not have moderate or severe exacerbation in the year prior to the study visit, (i.e. within the last 365 days before the study visit). Data related to history and details of exacerbations and ICS treatment, as well as data on current ICS treatment was obtained from medical charts.
  Moderate exacerbation: increase in, or new onset of, ≥ 2 respiratory symptoms (cough, sputum, dyspnea, wheezing, chest tightness) with ≥ 1 symptom lasting ≥ 3 days and leading the patient's attending physician to initiate treatment with systemic corticosteroids and/or antibiotics.
  Severe exacerbation: increase in or new onset of ≥ 2 respiratory symptoms (cough, sputum, dyspnoea, wheezing, chest tightness) with ≥ 1 symptom lasting ≥ 3 days and leading to patient's hospitalization.
Time Frame: 1 year prior to study visit, data collected at study visit (1 day).
Population: Patients in the FAS who were treated with ICS at study visit.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | COPD Patients Treated With ICS at Study Visit
Number analyzed (Participants) | 432
Percentage of participants | 62.5 [57.8 to 67.0]

2. Secondary Outcome: Percentage of Patients Currently on Inhaled CorticoSteroids (ICS) Who Have Had Moderate or Severe Exacerbation in the Year Prior to the Study Visit
Description: Percentage of patients currently on ICS who have had moderate or severe exacerbation in the year prior to the study visit, (i.e. within the last 365 days before the study visit). Data related to history and details of exacerbations and ICS treatment, as well as data on current ICS treatment was obtained from medical charts.
  Moderate exacerbation: increase in, or new onset of, ≥ 2 respiratory symptoms (cough, sputum, dyspnea, wheezing, chest tightness) with ≥ 1 symptom lasting ≥ 3 days and leading the patient's attending physician to initiate treatment with systemic corticosteroids and/or antibiotics.
  Severe exacerbation: increase in or new onset of ≥ 2 respiratory symptoms (cough, sputum, dyspnoea, wheezing, chest tightness) with ≥ 1 symptom lasting ≥ 3 days and leading to patient's hospitalization.
Time Frame: 1 year prior to study visit, data collected at study visit (1 day).
Population: Patients in the FAS who were treated with ICS at study visit.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | COPD Patients Treated With ICS at Study Visit
Number analyzed (Participants) | 432
Percentage of participants | 37.5 [32.9 to 42.3]

3. Secondary Outcome: Percentage of Patients Treated With Inhaled CorticoSteroids (ICS) at the Time of Study Visit With or Without Moderate or Severe Exacerbations, in the Previous 2 Years Before the Study Visit
Description: Percentage of patients with chronic obstructive pulmonary disease (COPD) treated with Inhaled CorticoSteroids (ICS) at the time of study visit with or without moderate or severe exacerbations, in the previous 2 years before the study visit. Data related to history and details of exacerbations and ICS treatment, as well as data on current ICS treatment was obtained from medical charts.
  Moderate exacerbation: increase in, or new onset of, ≥ 2 respiratory symptoms (cough, sputum, dyspnea, wheezing, chest tightness) with ≥ 1 symptom lasting ≥ 3 days and leading the patient's attending physician to initiate treatment with systemic corticosteroids and/or antibiotics.
  Severe exacerbation: increase in or new onset of ≥ 2 respiratory symptoms (cough, sputum, dyspnoea, wheezing, chest tightness) with ≥ 1 symptom lasting ≥ 3 days and leading to patient's hospitalization.
Time Frame: 2 years prior to study visit, data collected at study visit (1 day).
Population: Patients in the FAS who were treated with ICS at study visit.
Measure: Number; unit: Percentage of participants
Arm/Group | COPD Patients Treated With ICS at Study Visit
Number analyzed (Participants) | 432
Percentage of participants
  With moderate or severe exacerbations | 46.8
  Without moderate or severe exacerbations | 53.2

4. Secondary Outcome: Percentage of Patients Not Treated With Inhaled CorticoSteroids (ICS) at the Time of Study Visit With or Without Moderate or Severe Exacerbations, Both in the Previous 1 Year and Previous 2 Years Before the Study Visit
Description: Percentage of patients with chronic obstructive pulmonary disease (COPD) treated with Inhaled CorticoSteroids (ICS) at the time of study visit with or without moderate or serve exacerbations, both in the previous 1 year and previous 2 years before the study visit. Data related to history and details of exacerbations and ICS treatment, as well as data on current ICS treatment was obtained from medical charts.
  Moderate exacerbation: increase in, or new onset of, ≥ 2 respiratory symptoms (cough, sputum, dyspnea, wheezing, chest tightness) with ≥ 1 symptom lasting ≥ 3 days and leading the patient's attending physician to initiate treatment with systemic corticosteroids and/or antibiotics.
  Severe exacerbation: increase in or new onset of ≥ 2 respiratory symptoms (cough, sputum, dyspnoea, wheezing, chest tightness) with ≥ 1 symptom lasting ≥ 3 days and leading to patient's hospitalization.
Time Frame: 1 year and 2 years prior to study visit, data collected at study visit (1 day).
Population: Patients in the FAS who were not treated with ICS at study visit.
Measure: Number; unit: Percentage of participants
Arm/Group | COPD Patients Not Treated With ICS at Study Visit
Number analyzed (Participants) | 469
Percentage of participants
  1 year prior study visit: With moderate or severe exacerbations | 16.6
  1 year prior study visit: Without moderate or severe exacerbations | 83.4
  2 years prior study visit: With moderate or severe exacerbation | 22.8
  2 years prior study visit: Without moderate or severe exacerbations | 77.2

5. Secondary Outcome: Number of Moderate or Severe Exacerbations in Patients Treated With Inhaled Corticosteroids (ICS) at the Time of Study Visit, Both in Previous 1 Year and Previous 2 Years Before the Study Visit
Description: Number of moderate or severe exacerbations in chronic obstructive pulmonary disease (COPD) patients treated with ICS at the time of study visit, both in previous 1 year and previous 2 years before the study visit. Data related to history and details of exacerbations and ICS treatment, as well as data on current ICS treatment was obtained from medical charts.
  Moderate exacerbation: increase in, or new onset of, ≥ 2 respiratory symptoms (cough, sputum, dyspnea, wheezing, chest tightness) with ≥ 1 symptom lasting ≥ 3 days and leading the patient's attending physician to initiate treatment with systemic corticosteroids and/or antibiotics.
  Severe exacerbation: increase in or new onset of ≥ 2 respiratory symptoms (cough, sputum, dyspnoea, wheezing, chest tightness) with ≥ 1 symptom lasting ≥ 3 days and leading to patient's hospitalization.
Time Frame: 1 year and 2 years prior to study visit, data collected at study visit.
Population: Patients in the FAS who were treated with ICS at study visit.
Measure: Mean (Standard Deviation); unit: Exacerbations
Arm/Group | COPD Patients Treated With ICS at Study Visit
Number analyzed (Participants) | 432
Exacerbations
  1 year prior study visit | 0.72 (1.23)
  2 years prior to study visit | 1.27 (1.99)

6. Secondary Outcome: Number of Moderate or Severe Exacerbations in Patients Not Treated With Inhaled Corticosteroids (ICS) at the Time of Study Visit, Both in Previous 1 Year and Previous 2 Years Before the Study Visit
Description: Number of moderate or severe exacerbations in chronic obstructive pulmonary disease (COPD) patients not treated with ICS at the time of study visit, both in previous 1 year and previous 2 years before the study visit.Data related to history and details of exacerbations and ICS treatment, as well as data on current ICS treatment was obtained from medical charts.
  Moderate exacerbation: increase in, or new onset of, ≥ 2 respiratory symptoms (cough, sputum, dyspnea, wheezing, chest tightness) with ≥ 1 symptom lasting ≥ 3 days and leading the patient's attending physician to initiate treatment with systemic corticosteroids and/or antibiotics.
  Severe exacerbation: increase in or new onset of ≥ 2 respiratory symptoms (cough, sputum, dyspnoea, wheezing, chest tightness) with ≥ 1 symptom lasting ≥ 3 days and leading to patient's hospitalization.
Time Frame: 1 year and 2 years prior to study visit, data collected at study visit.
Population: Patients in the FAS who were not treated with ICS at study visit.
Measure: Mean (Standard Deviation); unit: Exacerbations
Arm/Group | COPD Patients Not Treated With ICS at Study Visit
Number analyzed (Participants) | 469
Exacerbations
  1 year prior study visit | 0.26 (0.77)
  2 years prior study visit | 0.43 (1.25)

7. Secondary Outcome: Percentage of Patients Using Rescue Medication
Description: Percentage of patients who used rescue medication (by type of rescue medication) in the last year and in the last two years. This percentage was calculated using as denominator the FAS set and was stratified by ICS treatment in the study visit.
  Data was obtained from medical charts.
  SABA: Short-acting beta2- agonists [*]: Salbutamol alone, terbutaline alone and salbutamol in combination (IPRATROPIUM BROMIDE /SALBUTAMOL) are included.
Time Frame: 1 year (last year) and 2 years (last 2 years) prior to study visit, data was collected at study visit (1 day).
Population: Full Analysis Set (FAS): Patients who provided informed consent and fulfilled all selection criteria.
Measure: Number; unit: Percentage of participants
Arm/Group | COPD Patients Not Treated With ICS at Study Visit | COPD Patients Treated With ICS at Study Visit
Number analyzed (Participants) | 469 | 432
Percentage of participants
  Last 2 years: Use of rescue medication (overall) | 43.9 | 65.7
  Last 2 years: Rescue Medication - SABA | 35.4 | 58.6
  Last 2 years: Rescue Medication - SABA[*] (including salbutamol in combinations) | 35.4 | 58.8
  Last 2 years: Rescue Medication - Others | 10.0 | 12.3
  Last 2 years: R03AC: Selective Beta-2-Adrenoreceptor Agonists | 35.6 | 58.6
  Last 2 years: R03BB: Anticholinergics | 9.2 | 10.9
  Last year: Use of rescue medication (overall) | 41.4 | 63.9
  Last year: Rescue medication - SABA | 33.0 | 56.9
  Last year: Rescue medication - SABA[*] (including salbutamol in combinations) | 33.0 | 57.2
  Last year: Rescue medication - Others | 9.6 | 11.3
  Last year: R03AC: Selective Beta-2-Adrenoreceptor Agonists | 33.0 | 56.9
  Last year: R03BB: Anticholinergics | 9.0 | 10.0

8. Secondary Outcome: Number of Patients With Adherence to Treatment Recommendations According Spanish COPD Guidelines (GesEPOC) 2017
Description: Number of patients with adherence to treatment recommendations according GesEPOC 2017 guidelines, stratified by risk and phenotypes.
  Adherence: Patients treated with Inhaled CorticoSteroids (ICS) that according to GesEPOC 2017 should had been treated with ICS; Patients not treated with ICS that according to GesEPOC 2017 should not had been treated with ICS.
  Non-adherence: Patients treated with ICS but according to GesEPOC 2017 should not have been treated with ICS; Patients not treated with ICS but according to GesEPOC 2017 should have been treated with ICS.
  Low risk: Patients with Forced Expiratory Volume in 1st second (FEV1) post bronchodilator ≥50% and Modified Medical Research Council (mMRC) (0-1-2) and with ≤1 moderate/severe exacerbation without hospitalization in the last year.
  High risk: Patients with FEV1 post bronchodilator <50% or mMRC (3-4) and ≥2 moderate/severe exacerbation or severe ≥1 in the last year. Current phenotype was assigned to high risk patients.
Time Frame: 1 year prior to study visit, data collected at study visit (1 day).
Population: Patients in the FAS with available type of risk and phenotype (n=877).
Measure: Count of Participants; unit: Participants
Arm/Group | COPD Patients Treated With ICS at Study Visit | COPD Patients Not Treated With ICS at Study Visit
Number analyzed (Participants) | 415 | 462
Participants
  Global: Adherence | 150 | 423
  Global: Non-Adherence | 265 | 39
  Low Risk: number analyzed (Participants) | 112 | 214
  Low Risk: Adherence | 0 | 214
  Low Risk: Non-Adherence | 112 | 0
  High Risk: number analyzed (Participants) | 303 | 248
  High Risk: Adherence | 150 | 209
  High Risk: Non-Adherence | 153 | 39

9. Secondary Outcome: Percentage of Patients With ICS-related Adverse Events
Description: Percentage of patients with adverse reactions commonly related to Inhaled CorticoSteroids (ICS), which were predefined in the eCRF and per protocol. In this sense, it could be the case of a patient reporting a commonly ICS-related adverse event, without current treatment with ICS at the time of the study visit. Data were obtained from medical charts. Results were reported for COPD patients overall (both arms combined), as the outcome is not related with the current ICS treatment of a patient.
Time Frame: 2 years prior to study visit, data collected at study visit (1 day).
Population: Full Analysis Set (FAS): Patients who provided informed consent and fulfilled all selection criteria.
Measure: Number; unit: Percentage of Participants
Groups:
- Patients With COPD - Overall: Patients with chronic obstructive pulmonary disease (COPD), with or without current treatment of Inhaled CorticoSteroids (ICS) at study visit.
Arm/Group | Patients With COPD - Overall
Number analyzed (Participants) | 901
Percentage of Participants | 1.55

10. Secondary Outcome: General Patient Profile - Body Mass Index (BMI)
Description: General patient profile for patients treated with inhaled corticosteroid (ICS) and patients not treated with ICS - Body Mass Index (BMI).
  Weight (in kg) and height (in cm) were collected in the electronic case report form (eCRF). Body Mass Index was calculated (with last measure available): BMI (kg/m^2) = weight (kg)/ height (m). BMI is categorized into 5 categories according to the World Health Organization (WHO):
  Underweight: BMI< 18.5 kg/m^2; Normal weight: 18.5 kg/m^2 ≤ BMI ≤ 25 kg/m^2; Overweight: 25 kg/m^2< BMI ≤ 30 kg/m^2; Obese: 30 kg/m^2 < BMI ≤ 35 kg/m^2; Severely Obese: BMI > 35 kg/m^2.
Time Frame: 2 years prior to study visit, data collected at study visit (1 day).
Population: Patients in the FAS with available data for this endpoint.
Measure: Mean (Standard Deviation); unit: Kg/m^2
Arm/Group | COPD Patients Treated With ICS at Study Visit | COPD Patients Not Treated With ICS at Study Visit
Number analyzed (Participants) | 407 | 446
Kg/m^2 | 28.38 (5.26) | 28.37 (5.11)

11. Secondary Outcome: General Patient Profile - Number of Patients by Smoking Habit
Description: General patient profile for patients treated with inhaled corticosteroids (ICS) and not treated with ICS. Number of patients by smoking habit (non-smoker, smoker, ex-smoker).
Time Frame: 2 years prior to study visit, data collected at study visit (1 day).
Population: Patients in the FAS with available data for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | COPD Patients Treated With ICS at Study Visit | COPD Patients Not Treated With ICS at Study Visit
Number analyzed (Participants) | 430 | 469
Participants
  Non-smoker | 36 | 42
  Smoker | 124 | 157
  Ex-smoker | 270 | 270

12. Secondary Outcome: General Patient Profile - Time Since Chronic Obstructive Pulmonary Disease (COPD) Diagnosis
Description: General patient profile for patients treated with inhaled corticosteroids (ICS) and not treated with ICS - time since COPD diagnosis.
  The year of the COPD diagnosis was collected in the electronic case report form (eCRF). The number of years since diagnosis was obtained as the difference between year of study visit and year of COPD diagnosis (+1).
Time Frame: Data collected at study visit.
Population: Full Analysis Set (FAS): Patients who provided informed consent and fulfilled all selection criteria.
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | COPD Patients Treated With ICS at Study Visit | COPD Patients Not Treated With ICS at Study Visit
Number analyzed (Participants) | 432 | 469
Years | 10.19 (6.10) | 8.93 (5.48)

13. Secondary Outcome: General Patient Profile - Number of Patients by Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2019 Spirometric Classification
Description: General patient profile for patients treated with inhaled corticosteroids (ICS) and not treated with ICS - Number of patients by GOLD 2019 spirometric classification. GOLD 2019 spirometric classification was auto-calculated according to the information recorded in the eCRF. While the protocol of the study planned to use GOLD 2017 guidelines, guideline updates were expected and it was planned to consider these updates for analysis purposes. For this reason, given that the GOLD 2019 guidelines were updated and effective, this guideline was used for auto-calculation. Spirometric data was collected from clinical records. To determine the severity of all subjects with COPD, patients were categorized into four levels based on their airflow limitation severity (based on post-bronchodilator FEV1 value): Gold 1 (mild): FEV1 (%) ≥ 80% predicted; Gold 2 (Moderate): 50% ≤ FEV1 (%) < 80% predicted; Gold 3 (Severe): 30% ≤ FEV1 (%) < 50% predicted; Gold 4 (Very serious): FEV1 (%) < 30% predicted.
Time Frame: 2 years prior to study visit, auto-calculated at study visit.
Population: Patients in the FAS with available data for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | COPD Patients Treated With ICS at Study Visit | COPD Patients Not Treated With ICS at Study Visit
Number analyzed (Participants) | 307 | 326
Participants
  Gold I - Mild | 57 | 85
  Gold II - Moderate | 164 | 194
  Gold III - Severe | 75 | 42
  Gold IV - Very Severe | 11 | 5

14. Secondary Outcome: General Patient Profile - Number of Patients by Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2019 Patient Groups
Description: General patient profile for patients treated with inhaled corticosteroids (ICS) and not treated with ICS - Number of patients by GOLD 2019 patient group (group A, group B, group C, group D).
  The GOLD 2019 patient group was auto-calculated according the information recorded in the eCRF.
  According to GOLD 2019 classification, four different types of patient groups were considered regarding their symptom burden and risk of exacerbation (exacerbations, Modified Medical Research Council (mMRC) and COPD Assessment Test (CAT) scores obtained from the eCRF):
  Group A: 0 or 1 exacerbations (not leading to hospital admission) and mMRC 0-1 and CAT < 10; Group B: 0 or 1 exacerbations (not leading to hospital admission), and mMRC ≥ 2 or CAT ≥ 10; Group C: ≥ 2 exacerbations or ≥ 1 exacerbation leading to hospital admission, and mMRC 0-1 and CAT < 10; Group D: ≥2 exacerbations or any ≥ 1 exacerbation leading to hospital admission, and mMRC ≥ 2 or CAT ≥ 10.
Time Frame: 2 years prior to study visit, auto-calculated at study visit.
Population: Full Analysis Set: Patients who provided informed consent and fulfilled all selection criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | COPD Patients Treated With ICS at Study Visit | COPD Patients Not Treated With ICS at Study Visit
Number analyzed (Participants) | 432 | 469
Participants
  Group A | 39 | 54
  Group B | 224 | 330
  Group C | 3 | 6
  Group D | 166 | 79

15. Secondary Outcome: General Patient Profile - Body Mass Index, Airflow Obstruction, Dyspnea and Exacerbations (BODEx) Index
Description: General patient profile for patients treated with inhaled corticosteroids (ICS) and patients not treated with ICS - BODEx index. The BODEx index is used to predict the mortality rate from chronic obstructive pulmonary disease (COPD). The BODEx index was auto-calculated according the information recorded in the eCRF.
  It includes the body mass index (BMI), the degree of dyspnea measured with the mMRC (Modified Medical Research Council) scale, the pulmonary function measured with the FEV1 (%) post-bronchodilation and the number of severe exacerbations (only visits to hospital emergencies and admissions are included).
  For each item, a score (0-3) is calculated. BODEx index is obtained as the sum of the scores of all items.
  The index ranges from 0 to 9, with a higher index indicating a higher risk of death.
Time Frame: 2 years prior to study visit, auto-calculated at study visit (1 day).
Population: Patients in the FAS with available data for this endpoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | COPD Patients Treated With ICS at Study Visit | COPD Patients Not Treated With ICS at Study Visit
Number analyzed (Participants) | 297 | 315
Score on a scale | 1.93 (1.72) | 1.15 (1.21)

16. Secondary Outcome: General Patient Profile - COPD Assessment Test (CAT) Score
Description: General patient profile for patients treated with inhaled corticosteroids (ICS) and patients not treated with ICS - CAT score.
  The CAT score was obtained from the sum of 8 items (cough, mucus, chest pressure, dyspnea, limitation in domestic activities, social limitation, sleep, energy). Each item ranging from 0 (no symptoms) to 5 points (highest symptoms). To obtain a valid score, no missing values or missing answers were allowed. The total score was obtained as the sum of the scores of all items, ranging from 0 - 40.
  The score was grouped into two categories:
  CAT <10: Low impact of COPD (Most days are good, the illness prevents the patient from doing one or two things he or she would like, coughing several days a week);CAT ≥10: Medium / high impact of COPD in the patient.
Time Frame: Data measured at study visit.
Population: Full Analysis Set: Patients who provided informed consent and fulfilled all selection criteria.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | COPD Patients Treated With ICS at Study Visit | COPD Patients Not Treated With ICS at Study Visit
Number analyzed (Participants) | 432 | 469
Score on a scale | 16.06 (8.03) | 12.96 (7.25)

17. Secondary Outcome: General Patient Profile - Number of Patients by Modified Medical Research Council (mMRC) Score
Description: General patient profile for patients treated with inhaled corticosteroids (ICS) and patients not treated with ICS - mMRC score.
  The mMRC score was used to assess severity of breathlessness in chronic obstructive pulmonary disease (COPD) patients.
  Patients were asked to answer the breathlessness scale (Mmrc), a single item (0-4) scale assessing current level of dyspnea. The mMRC comprised of five statements that describe almost the entire range of respiratory disability from none (grade 0) to almost complete incapacity (grade 4). A lower (higher) grade is considered a better (worse) outcome.
  Grade 0: None severity Grade 1: Mild severity Grade 2: Moderate severity Grade 3: Severe severity Grade 4: Very severe severity
Time Frame: Data measured at study visit.
Population: Full Analysis Set: Patients who provided informed consent and fulfilled all selection criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | COPD Patients Treated With ICS at Study Visit | COPD Patients Not Treated With ICS at Study Visit
Number analyzed (Participants) | 432 | 469
Participants
  Grade 0 | 58 | 93
  Grade 1 | 142 | 199
  Grade 2 | 133 | 130
  Grade 3 | 70 | 44
  Grade 4 | 29 | 3

18. Secondary Outcome: General Patient Profile - Number of Patients by Level of Eosinophils
Description: General patient profile for patients treated with inhaled corticosteroids (ICS) and patients not treated with ICS - level of eosinophils. Reported is the number of patients by category (low number of eosinophils, high number of eosinophils). Data is obtained from medical charts. Eosinophils were collected in cells per microliter (µl) and the categories are defined as followed:
  Low number of eosinophils: < 300 cel/µl; High number of eosinophils: ≥ 300 cel/µl.
Time Frame: 2 years prior to study visit, data collected at study visit (1 day).
Population: Patients in the FAS with available data for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | COPD Patients Treated With ICS at Study Visit | COPD Patients Not Treated With ICS at Study Visit
Number analyzed (Participants) | 304 | 328
Participants
  Low number of eosinophils | 208 | 242
  High number of eosinophils | 96 | 86

19. Secondary Outcome: General Patient Profile - Number of Patients by Current Chronic Obstructive Pulmonary Disease (COPD) Treatment
Description: General patient profile for patients treated with inhaled corticosteroid (ICS) and patients not treated with ICS: Current COPD treatment (treatment patterns for COPD) according to current treatment on ICS. Reported is the number of patients by current COPD treatment. Data is obtained from medical charts.
  LABA: Long-Acting Beta2-Agonist; LAMA: Long-Acting Muscarinic Antagonist; SABA: Short-acting beta2- agonists; SAMA: Short-acting muscarinic antagonist.
Time Frame: 2 years prior to study visit, data collected at study visit.
Population: Full Analysis Set: Patients who provided informed consent and fulfilled all selection criteria.
Measure: Count of Participants; unit: Participants
Groups:
- COPD Patients Not Treated With ICS at Study Visit: Patients with chronic obstructive pulmonary disease (COPD) currently (at study visit) treated with Inhaled CorticoSteroids (ICS).
Arm/Group | COPD Patients Treated With ICS at Study Visit | COPD Patients Not Treated With ICS at Study Visit
Number analyzed (Participants) | 432 | 469
Participants
  Without treatment | 0 | 46
  SABA alone | 0 | 6
  SAMA alone | 0 | 5
  SABA + SAMA | 0 | 0
  LABA alone | 0 | 3
  LAMA alone | 0 | 93
  ICS alone | 5 | 0
  LABA + LAMA | 0 | 316
  LABA + ICS | 106 | 0
  LAMA + ICS | 4 | 0
  LABA + LAMA + ICS | 317 | 0

ADVERSE EVENTS:
Time Frame: Within 2 years prior to the study visit, up to 2 years.
Description: The study design is of non-interventional nature and the study is conducted within the conditions of the approved marketing authorizations. As no investigational product was used, but patients could have been treated with BI drugs, adverse events were reported on the safety analysis set, which included all enrolled patients treated with at least on dose of SPIOLTO®, STRIVERDI®, SPIRIVA® or ATROVENT® during the study period. Adverse events were reported as single arm align with the study design.
Groups:
- COPD Patients Treated or Not Treated With ICS at Study Visit: Patients with chronic obstructive pulmonary disease (COPD) currently (at study visit) treated or not treated with Inhaled CorticoSteroids (ICS).
Arm/Group | COPD Patients Treated or Not Treated With ICS at Study Visit
All-Cause Mortality (participants affected / at risk) | 0/441
Serious Adverse Events (participants affected / at risk) | 0/441
Other Adverse Events (participants affected / at risk) | 0/441

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-09-19): https://cdn.clinicaltrials.gov/large-docs/77/NCT03611777/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT03611777/SAP_002.pdf